CLINICAL TRIAL: NCT01705470
Title: Furosemide Treatment Before Blood Transfusion in Patients With Systolic Dysfunction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the medical center, no replacement assigned
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHERLOCK
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Anemia Treatment Among Patients Suffering From Left Ventricular Systolic Dysfunction
Keywords: Furosemide; Anemia; LV dysfunction; blood transfusion
MeSH Terms: conditions — Anemia; Ventricular Dysfunction, Left | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm1 (Experimental): will receive 60 mg (6 ml) of intra-venous furosemide before administration of the blood transfusion (250-300 ml of packed cells).
  Interventions: Drug: furosemide
- arm2 (Experimental): will receive 6 ml of normal saline (NaCl 0.9%) before administration of the blood transfusion (250-300 ml of packed cells).
  Interventions: Drug: placebo normal saline

INTERVENTIONS:
Drug: furosemide
  Arms: arm1
Drug: placebo normal saline
  Arms: arm2

SUMMARY:
The study Objective is to assess the clinical and echocardiographic changes of patients with systolic dysfunction receiving blood transfusion, with or without prior treatment with furosemide

DETAILED DESCRIPTION:
More than 4 million patients receive a blood transfusion each year in the United States, many of them suffer from congestive heart failure. The reported prevalence of anemia in CHF is unknown, ranges widely from 4% to 70%, due to a lack of an established, consistent definition of anemia in CHF.

Treating CHF patients with furosemide prior to blood transfusion became a common practice, even though no randomize clinical trial had examine this issue. Nand et al. measured the pulmonary capillary wedge pressures in 20 adults with chronic severe anemia (Hg <6 mg/dl) and no systemic disease before and after transfusion of 700ml of whole blood. Ten of these patients were treated with furosemide (40 mg intra-venous) immediately prior the transfusion. The PCWP had increased significantly among patient who did not receive the furosemide and decreased by 3.75% among patients in the furosemide group, although this change was not was statistically significant. In another study, the same group of Nand et al. measured the PCWP among 40 chronic anemia patients receiving blood transfusion. None of the patients suffered from cardiopulmonary disease. The patients were randomly divided into 4 groups: the difference between the first 3 groups was the speed of the transfusion (2 ml/min, 5 ml/min and 10 ml/min). The fourth group patients were treated with 40 mg of furosemide before the transfusion was given in a rate of 5 ml/min. The PCWP increased significantly in the first 3 groups, with the rise being proportionately greater with faster transfusions (15.8, 20.9 and 32.2% in groups A, B and C, respectively). In the furosemide group, however, the PCWP decreased significantly by 21.7%.

ELIGIBILITY:
Inclusion Criteria:

* Subject is over 18 years old.
* Documented ejection function equal to or over 40% in prior tests
* The treating physician decided to treat the patient with packed cell

Exclusion Criteria:

* Known hypersensitivity to furosemide.
* Calculated creatinine clearance over 20% (by MDRD)
* Past adverse reaction to blood product.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Diastolic echocardiographic changes following blood transfusion, with or without Furosemide treatment | Within 4 hours from receiving the blood transfusion
  Diastolic echocardiographic variables, including Ea, E to Ea ratio, E to A ratio, and Pulmonary vein flow velocities, following blood transfusion, with or without Furosemide treatment

SECONDARY OUTCOMES:
clinical outcome following blood transfusion, with or without Furosemide treatment | Within 4 hours from receiving the blood transfusion
  clinical outcome variables following blood transfusion, with or without Furosemide treatment, including the respiratory rate and oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Edo Birati, MD, Principal Investigator — Tel Aviv MC

IPD SHARING:
Plan to Share IPD: No